CLINICAL TRIAL: NCT05863988
Title: Effects Of Functional Electrical Stimulation Versus Upper Limb Loading Exercises on Grip Strength,Dexterity and Function in Patients With Spinal Cord Injury
Brief Title: FES and Upper Limb Loading Exercises Outcome Comparison on Hand Function in Spinal Cord Injury Patients
Acronym: OCONHAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/LHR/23/0214 Aroosa
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Spinal Cord Injuries
Keywords: Dexterity,Functional Electrical Stimulation,Hand Function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Electrical Stimulation &upper limb loading exercises (Active Comparator): The group A Will receive functional electrical stimulation and conservative treatment 30-45 min session 5 days per week for 8 weeks.
  Interventions: Other: Functional Electrical Stimulation
- Functional Electrical Stimulation & Upper Limb Loading Exercises (Active Comparator): The group B will receive upper limb loading exercises and conservative treatment 30-45 min session 5 days per week for 8 weeks.
  Interventions: Other: Upper Limb Loading Exercises

INTERVENTIONS:
Other: Functional Electrical Stimulation — The group A will receive functional electrical stimulation 30-45 min session 5 days per week for 8 weeks.
  Arms: Functional Electrical Stimulation &upper limb loading exercises
Other: Upper Limb Loading Exercises — The group B will receive Upper Limb Loading Exercises 30-45 min session 5 days per week for 8 weeks.
  Arms: Functional Electrical Stimulation & Upper Limb Loading Exercises

SUMMARY:
This study is conducted to assess the effectiveness of functional electrical stimulation Vs limb loading exercises on hand grip strength,dexterity and function in patients with subacute cervical spinal cord injury.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is based on the concept that rehabilitative training recruits neuronal systems spinal cord injury that remain intact after the injury to take over the impaired function.Working in the field of rehabilitation of the spinal cord injured, presents many challenges. Every patient presents a new and specific challenge. The tetraplegics more so than the paraplegics as the result of loss of active function of their upper extremities in addition to loss of function in the trunk and lower extremities. This study will be conducted to assess the effects of functional electrical stimulation versus limb loading exercises on hand grip strength,dexterity and function in patients with subacute spinal cord injury.

trength,dexterity and function in patients with subacute spinal cord injury. The study will be randomized clinical trial. Participants will be randomly allocated in to two groups each group will have ten participants.. This study will be conducted in two Hospitals in Punjab pakistan. The group A Will receive functional electrical stimulation .The group B will receive upper limb loading exercises .Both groups will be given 30-45 min session 5 days per week for 8 weeks. The outcomes will be measured before and after giving treatment by using modified Action Research Arm Test (ARAT),Hand held dynamometry , Nine-Hole Peg Test (9HPT). The results will be calculated by using SPSS 23 version . Statistical tests will be applied according to the normality of the data either it will be parametric or non-parametric.

ELIGIBILITY:
Inclusion Criteria:

* Patients with incomplete SCI at neurological level C5-T1 in subacute stage.
* Medically stable
* Able to tolerate the Functional Electrical stimulation without sustained autonomic dysreflexia
* A score greater than 16 in mini-mental test

Exclusion Criteria:

* Patients taking long term steroids
* patient having pre-existing injury on upper limb or hand
* Patients have had Previous participation in experimental trial for spinal cord injury
* Patients using Currently cardioactive medications
* Individuals who has had Tendon transfers, implanted devices bladder stimulation, chronic intrathecal infusions
* Individuals with Bleeding disorders.
* Amputation of any digit on target hand

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-10-18 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Modified Action Research Arm Test | 8th week
  The ARAT has excellent reliability and low ceiling effects. It consists of 4 subtests, including grasp, grip, pinch, and gross movement. All tasks were scored on a 4-point scale from 0 to 3, where 0 reflects poor hand function and 3 reflects good hand function (maximum score, 57).
Hand Held Dynamometry | 8th week
  A small portable device is held by the examiner and placed against the patient's limb .during a maximal isometric contraction. The device can be used to test hand muscle strength efficiently
9 peg hole test | 8th week
  Nine-Hole Peg Test is administered by asking the client to take the pegs from a container, one by one, and place them into holes on the board as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container.. The number of seconds it takes for the patient to complete the test.

CONTACTS AND LOCATIONS:
Overall Officials: Hira jabeen, MS NMPT, Principal Investigator — Riphah International University
Locations (1):
- Bahawal Victoria Hospital Bahawalpur, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson KD. Targeting recovery: priorities of the spinal cord-injured population. J Neurotrauma. 2004 Oct;21(10):1371-83. doi: 10.1089/neu.2004.21.1371. PMID 15672628
- [Background] Beekhuizen KS, Field-Fote EC. Massed practice versus massed practice with stimulation: effects on upper extremity function and cortical plasticity in individuals with incomplete cervical spinal cord injury. Neurorehabil Neural Repair. 2005 Mar;19(1):33-45. doi: 10.1177/1545968305274517. PMID 15673842
- [Background] Hilton BJ, Anenberg E, Harrison TC, Boyd JD, Murphy TH, Tetzlaff W. Re-Establishment of Cortical Motor Output Maps and Spontaneous Functional Recovery via Spared Dorsolaterally Projecting Corticospinal Neurons after Dorsal Column Spinal Cord Injury in Adult Mice. J Neurosci. 2016 Apr 6;36(14):4080-92. doi: 10.1523/JNEUROSCI.3386-15.2016. PMID 27053214